CLINICAL TRIAL: NCT04067921
Title: Platform for Clinical Trials in Nutrition and Health
Acronym: GENYALPlatform
Status: Active, not recruiting | Type: Observational
Sponsor: IMDEA Food (Other)
Responsible Party: Sponsor
Other Study IDs: CEI 27-666
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Precision Nutrition; Nutritional Genetics; Nutritional Genomics; Polymorphisms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the known link between dietary patterns and disease, it has been observed that the specific response of each individual to dietary components highly varied, and this may limit the impact of the nutritional interventions to improve public health. These observations provided the basis to the development of the Nutritional Genomics at the beginning of the 90s, which main goal was to study the interaction between dietary factors and the genome that modulate phenotypic expression. From this idea, in the recent years, Precision Nutrition has been emerged as a therapeutic approach that takes into account all individual's characteristics to develop targeted nutritional advices. The main goal of Precision Nutrition is to maintain or improve health by using genetics, phenotypic, clinical, dietary and other information to provide more precise and more efficacious personalized healthy eating advice and to motivate appropriate dietary changes. However, all the genotype-dependent advice must be based on scientific evidence. Most of the available evidence in support of personalized nutrition has come from observational studies with risk factors as outcomes, and it was needed randomized controlled trials using clinical endpoints to ratify these results.

The main objective of the Platform for Clinical Trials in Nutrition and Health (GENYAL) is to contribute to Precision Nutrition Research by the construction, for the first time, of a human gene and phenotype database to be used in: 1) The evaluation of the efficacy of different foods, functional foods and bioactive compounds capsules on general population and by genotypes and 2) The performance of nutritional genetics and nutrigenomics studies. For that purposes, GENYAL has a permanent recruitment of volunteers, which are phenotypically and genotypically characterized, and give consent to be contacted to perform clinical trials and nutritional intervention studies. Therefore, GENYAL may help to increase the existing knowledge for moving along to Nutritional Genomics research to its practical application in Precision Nutrition; contributing in the improvement in health and disease prevention through dietary recommendations based on the genome.

ELIGIBILITY:
Inclusion Criteria:

* Free-living adults aged from 18 to 70 years that give written informed consent to be contacted to perform clinical trials and nutritional intervention studies.

Exclusion Criteria:

* Suffering from any serious illness (kidney or liver diseases or other condition that affects lifestyle or diet).
* Presenting dementia or impaired cognitive function
* Being pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Free-living adults aged from 18 to 70 years and residents of Spain.
Sampling Method: Non-Probability Sample
Enrollment: 1963 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Genotypic characterization. | Baseline.
  Genomic DNA is isolated from a blood sample. Genotyping was performed using the QuantStudio 12 K Flex Real-Time PCR System (Life Technologies Inc., Carlsbad, CA) with a TaqMan OpenArray plates.

SECONDARY OUTCOMES:
Changes in total daily energy intake (TEI). | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the TEI (kcal) of the sample.
Changes in macronutrients intake. | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the following variables:
  * Carbohydrates (grams per day and percentage of the TEI).
  * Proteins (grams per day and percentage of the TEI).
  * Lipids (grams per day and percentage of the TEI).
Changes in fatty acids intake. | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the saturated, unsaturated and polyunsaturated fatty acids intake (grams per day and percentage of the TEI).
Changes in cholesterol intake. | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the cholesterol intake (milligrams per day).
Changes in fiber intake. | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the fiber intake (grams per day).
Changes in sugar intake. | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the sugar intake (grams per day and percentage of the TEI).
Changes in micronutrients intake. | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the intake (grams, milligrams or micrograms, as the case may be) of the following variables:
  * Minerals: Ca, P, Mg, Fe, Zn, I, F, Se.
  * Vitamins: A, D, E, K, B1, B2, B5, B6, B12, biotin, niacin, folate.
Changes in nutritional quality of diet: Healthy Eating Index | At the beginning and before 12 months.
  Dietary intake is collected using a 72-hour food and drink record validated for the Spanish population. The DIAL software (Alce Ingeniería) is used to evaluate the nutritional quality of diet according to the Healthy Eating Index (Kennedy et al, 1995).
Changes in height. | At the beginning and before 12 months.
  This anthropometric measure (cm) is taken using a Leicester stadiometer (Biological Medical Technology SL, Barcelona, Spain) by trained nutritionists according to standardized procedures.
Changes in body composition: fat and lean mass. | At the beginning and before 12 months.
  Fat mass (%) and lean mass (%) are evaluated using a BF511 Body Composition Monitor (Omron Healthcare Co. Ltd., Kyoto, Japan).
Changes in weight. | At the beginning and before 12 months.
  Weight (kg) is evaluated using a BF511 Body Composition Monitor (Omron Healthcare Co. Ltd., Kyoto, Japan).
Changes in body mass index (BMI). | At the beginning and before 12 months.
  BMI (kg/m^2) is calculated according to the Quetelet Index ((Weight (kg))/〖Height (m)〗^2 ).
Changes in waist circumference. | At the beginning and before 12 months.
  Waist circumference (cm) is measured using a Seca 201 nonelastic tape (Quirumed, Valencia, Spain).
Changes in systolic (SBP) and diastolic blood pressure (DBP). | At the beginning and before 12 months.
  Both are measured using a Model M3 Automatic Digital Blood Pressure Monitor (Omron Healthcare Co. Ltd., Kyoto, Japan), according to standardized procedures.
Changes in physical activity pattern according to the Minnesota Leisure Time Physical Activity Questionnaire (MLTPAQ). | At the beginning and before 12 months.
  The validated Spanish version of the MLTPAQ is used to quantitatively measure the average physical activity practice (kcal/day) by the volunteers. Based on the Compendium of physical activities (PA), Energy Expenditure in Physical Activity (EEPA) is estimated as follows: EEPA = I x N x T; where "I" is the degree of intensity for each physical activity in kcal/min; "N", the number of times that physical activity is developed; and "T", the time in minutes spent in each session.
  The MLTPAQ is administered to assess the quality of PA according to their intensity code: low (intensity code of <=4 kcal/min), moderate (4.5-5.5 kcal/min) and high (>=6 kcal/min).
Changes in physical activity pattern according to the International Physical Activity Questionnaire (IPAQ). | At the beginning and before 12 months.
  Physical activity (PA) is assessed using the validated Spanish version of the IPAQ.
  The continuous score is expressed as metabolic equivalents (MET)-min per week: MET level x minutes of activity x events per week.
  The pattern of PA is classified into 3 categories in accordance with the intensity:
  * Low: the lowest level of physical activity.
  * Moderate: any one of the following criteria: >=3 days of vigorous activity of at least 20 min/day or >=5 days of moderate-intensity activity or walking of at least 30 min/ day or >=5 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-min/week.
  * High: any one of the following criteria: vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-min/week or >=7 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-min/week.
Number of participants with changes in lipid profile. | At the beginning and before 12 months.
  The following lipid parameters will be taking into account:
  * Triglycerides (TG)
  * Total Cholesterol (CT)
  * Low Density Lipoprotein (LDL)
  * Very Low Density Lipoprotein (VLDL)
  * High Density Lipoprotein (HDL)
  * CT/HDL ratio
  * LDL/HDL ratio
  * TG/HDL ratio
  * Apolipoprotein B100
  * Apolipoprotein E
  * Plasma free fatty acids (FFAs)
Number of participants with changes in glycemic profile. | At the beginning and before 12 months.
  The following glycemic parameters will be taking into account:
  * Glycemia
  * Insulin
  * Homeostasis Model Assessment (HOMA)
Number of participants with changes in biochemical parameters. | At the beginning and before 12 months.
  The following biochemical parameters will be taking into account:
  * LDL-ox
  * 8-iso PGF2α
Number of participants with changes in biochemical parameters associated with inflammation. | At the beginning and before 12 months.
  The following parameters will be taking into account:
  * PCRu
  * TNFα
  * IL1β
  * VCAM1
  * ICAM
  * TXB2
Number of participants with changes in blood clotting and endothelial function. | At the beginning and before 12 months.
  The following parameters will be taking into account:
  * PAI I
  * Fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ramírez, PhD, Study Director — IMDEA Food; Guillermo Reglero, Prof. PhD, Study Director — IMDEA Food; Viviana Loria-Kohen, PhD, Principal Investigator — IMDEA Food
Locations (1):
- IMDEA Food, Madrid, Spain

REFERENCES:
- [Derived] Camblor Murube M, Borregon-Rivilla E, Colmenarejo G, Aguilar-Aguilar E, Martinez JA, Ramirez De Molina A, Reglero G, Loria-Kohen V. Polymorphism of CLOCK Gene rs3749474 as a Modulator of the Circadian Evening Carbohydrate Intake Impact on Nutritional Status in an Adult Sample. Nutrients. 2020 Apr 19;12(4):1142. doi: 10.3390/nu12041142. PMID 32325849